CLINICAL TRIAL: NCT03457623
Title: Medico-economic Evaluation of a "IsereADOM" Package of Services Versus Conventional Health and Social Monitoring, in the Care of a Population of People With Heart Failure in Isère.
Brief Title: Batch n ° 2 of the Public Market Evaluation "Medico-economic Demonstrator IsereADOM"
Acronym: CardIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 38RC16.045
Record Dates: First submitted 2018-02-28; First posted 2018-03-07 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Innovative supported (Experimental): In addition to usual care, patients benefit from connected tools (overpoise, sphygmomanometer...), physical activity, a strong accompaniment with a referent person
  Interventions: Other: Innovative Supported
- conventional supported (No Intervention): Patients benefit from usual care

INTERVENTIONS:
Other: Innovative Supported — addition of connected tools and stronger accompaniment to improve quality of life
  Arms: Innovative supported

SUMMARY:
The goal of this study is to evaluate the health and social benefit of innovative management - IsereADOM - versus conventional follow-up in patients with heart failure.

There is a medico-economic goal too, is to perform a cost-utility analysis of the service bundle (IsereADOM) versus conventional 6-month community-based follow-up in a population with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with heart failure confirmed by a cardiologist ;
* Patient with functional NYHA II, III, IV staining ;
* Patient domiciled in the department of Isère ;
* Patient who can be followed regularly for 6 months ;
* Patient who can benefit from RESIC-type health education ;
* Presence of a caregiver referent of proximity (family or other) according to appreciation of the investigating doctor in case of cognitive disorders ;
* Patient affiliated with social security or beneficiary of such a scheme ;
* Patient able to read, write and understand French ;
* Patient having signed informed consent to participate.

Exclusion Criteria:

* Patient with peritoneal dialysis or haemofiltration ;
* Patient with severe co-morbidity with poor short-term prognosis: mortality < 6 months ;
* Patient with future surgical etiologic treatment: prosthetic valve, revascularization procedure, TAVI or MITRACLIP ;
* Patient residing in a nursing home or institution for dependent person ;
* Persons referred to in Articles L1121-5 to L1121-8 of the CSP (corresponds to all persons protected: pregnant woman, parturient, mother who is breastfeeding, person deprived of liberty by judicial or administrative decision, person subject of a legal protection measure).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
the effectiveness of a service package compared to conventional follow-up in people with heart failure. | 6 months
  The outcome measure is the number of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Muriel SALVAT, MD, Principal Investigator — CHU Grenoble Alpes
Locations (2):
- France (2):
  - Groupe Hospitalier Mutualiste, Grenoble
  - CHU Grenoble-Alpes, Grenoble

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mathers CD, Loncar D. Projections of global mortality and burden of disease from 2002 to 2030. PLoS Med. 2006 Nov;3(11):e442. doi: 10.1371/journal.pmed.0030442. PMID 17132052
- [Background] Desai AS, Stevenson LW. Rehospitalization for heart failure: predict or prevent? Circulation. 2012 Jul 24;126(4):501-6. doi: 10.1161/CIRCULATIONAHA.112.125435. No abstract available. PMID 22825412
- [Background] McMurray JJ, Adamopoulos S, Anker SD, Auricchio A, Bohm M, Dickstein K, Falk V, Filippatos G, Fonseca C, Gomez-Sanchez MA, Jaarsma T, Kober L, Lip GY, Maggioni AP, Parkhomenko A, Pieske BM, Popescu BA, Ronnevik PK, Rutten FH, Schwitter J, Seferovic P, Stepinska J, Trindade PT, Voors AA, Zannad F, Zeiher A; Task Force for the Diagnosis and Treatment of Acute and Chronic Heart Failure 2012 of the European Society of Cardiology; Bax JJ, Baumgartner H, Ceconi C, Dean V, Deaton C, Fagard R, Funck-Brentano C, Hasdai D, Hoes A, Kirchhof P, Knuuti J, Kolh P, McDonagh T, Moulin C, Popescu BA, Reiner Z, Sechtem U, Sirnes PA, Tendera M, Torbicki A, Vahanian A, Windecker S, McDonagh T, Sechtem U, Bonet LA, Avraamides P, Ben Lamin HA, Brignole M, Coca A, Cowburn P, Dargie H, Elliott P, Flachskampf FA, Guida GF, Hardman S, Iung B, Merkely B, Mueller C, Nanas JN, Nielsen OW, Orn S, Parissis JT, Ponikowski P; ESC Committee for Practice Guidelines. ESC guidelines for the diagnosis and treatment of acute and chronic heart failure 2012: The Task Force for the Diagnosis and Treatment of Acute and Chronic Heart Failure 2012 of the European Society of Cardiology. Developed in collaboration with the Heart Failure Association (HFA) of the ESC. Eur J Heart Fail. 2012 Aug;14(8):803-69. doi: 10.1093/eurjhf/hfs105. No abstract available. PMID 22828712
- [Background] Desai AS. The three-phase terrain of heart failure readmissions. Circ Heart Fail. 2012 Jul 1;5(4):398-400. doi: 10.1161/CIRCHEARTFAILURE.112.968735. No abstract available. PMID 22811548
- [Background] Takeda A, Taylor SJ, Taylor RS, Khan F, Krum H, Underwood M. Clinical service organisation for heart failure. Cochrane Database Syst Rev. 2012 Sep 12;(9):CD002752. doi: 10.1002/14651858.CD002752.pub3. PMID 22972058
- [Background] Krumholz HM, Merrill AR, Schone EM, Schreiner GC, Chen J, Bradley EH, Wang Y, Wang Y, Lin Z, Straube BM, Rapp MT, Normand SL, Drye EE. Patterns of hospital performance in acute myocardial infarction and heart failure 30-day mortality and readmission. Circ Cardiovasc Qual Outcomes. 2009 Sep;2(5):407-13. doi: 10.1161/CIRCOUTCOMES.109.883256. Epub 2009 Jul 9. PMID 20031870
- [Background] Powell LH, Calvin JE Jr, Richardson D, Janssen I, Mendes de Leon CF, Flynn KJ, Grady KL, Rucker-Whitaker CS, Eaton C, Avery E; HART Investigators. Self-management counseling in patients with heart failure: the heart failure adherence and retention randomized behavioral trial. JAMA. 2010 Sep 22;304(12):1331-8. doi: 10.1001/jama.2010.1362. PMID 20858878
- [Background] Manca A, Hawkins N, Sculpher MJ. Estimating mean QALYs in trial-based cost-effectiveness analysis: the importance of controlling for baseline utility. Health Econ. 2005 May;14(5):487-96. doi: 10.1002/hec.944. PMID 15497198